CLINICAL TRIAL: NCT04875533
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, THIRD-PARTY-UNBLINDED TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN PNEUMOCOCCAL VACCINE-NAÏVE ADULTS 60 YEARS OF AGE AND OLDER IN JAPAN, KOREA, AND TAIWAN
Brief Title: 20-valent Pneumococcal Conjugate Vaccine Safety and Immunogenicity Study in Pneumococcal Vaccine-Naïve Adults 60 Years of Age and Older in Japan, Korea, and Taiwan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B7471009
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — Sodium Chloride; 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 20vPnC/Saline (Experimental): 20vPnC and saline
  Interventions: Biological: 20vPnC; Other: Saline
- 13vPnC/PPSV23 (Active Comparator): 13vPnC and PPSV23
  Interventions: Biological: 13vPnC; Biological: PPSV23

INTERVENTIONS:
Biological: 20vPnC — 20vPnC
  Arms: 20vPnC/Saline
Other: Saline — Saline
  Arms: 20vPnC/Saline
Biological: 13vPnC — Pneumococcal conjugate vaccine
  Arms: 13vPnC/PPSV23
Biological: PPSV23 — Pneumococcal polysaccharide vaccine
  Other Names: Pneumovax 23
  Arms: 13vPnC/PPSV23

SUMMARY:
A phase 3, randomized, double-blind trial to evaluate the safety and immunogenicity of a 20-valent pneumococcal conjugate vaccine in pneumococcal vaccine-naïve adults 60 years of age and older in Japan, Korea, and Taiwan

ELIGIBILITY:
Inclusion criteria:

* Male or female participants 60 years of age and older at the time of consent.
* Adults determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study, including adults with preexisting stable disease, defined as disease not requiring significant change in therapy in the previous 6 weeks or hospitalization for worsening disease within 12 weeks before receipt of study intervention. (For adults 60 through 64 years of age to be enrolled at Japan sites: Participants must have a preexisting chronic stable disease with an elevated risk for pneumococcal disease.)

Exclusion criteria:

* History of microbiologically proven invasive disease caused by S pneumoniae.
* Serious chronic disorder, including metastatic malignancy, severe COPD requiring supplemental oxygen, end-stage renal disease with or without dialysis, cirrhosis of the liver, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
* Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt through study participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1425 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (28):
- Japan (10):
  - Seishinkai Inoue Hospital, Itoshima, Fukuoka
  - Women's Clinic LUNA NEXT STAGE, Naka-ku, Yokohama-Shi, Kanagawa
  - Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - P-one Clinic, Keikokai Medical Corporation, Hachioji-shi, Tokyo
  - Hillside Clinic Jingumae, Shibuya-ku, Tokyo
  - Medical Corporation Heishinkai ToCROM Clinic, Shinjuku-ku, Tokyo
  - SOUSEIKAI PS Clinic, Fukuoka
- South Korea (12):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University Hospital, Daegu
  - Inha University Hospital, Incheon
  - Severance Hospital, Yonsei University Health System, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Asan medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
- Taiwan (6):
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Haranaka M, Young Song J, Huang KC, de Solom R, Yamaji M, McElwee K, Kline M, Aizawa M, Peng Y, Scully I, Kogawara O, Gruber WC, Scott DA, Watson W. A phase 3 randomized trial of the safety and immunogenicity of 20-valent pneumococcal conjugate vaccine in adults >/= 60 years of age in Japan, South Korea, and Taiwan. Vaccine. 2024 Feb 15;42(5):1071-1077. doi: 10.1016/j.vaccine.2024.01.004. Epub 2024 Jan 23. PMID 38267330
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants 60 years of age and above were recruited into this study to received either Pneumococcal Conjugate Vaccine (20vPnC)/saline or 13-valent pneumococcal conjugate vaccine (13vPnC)/23-valent pneumococcal polysaccharide vaccine (PPSV23).
Pre-assignment Details: A total of 1425 participants were randomized to receive either 20vPnC/saline (713 participants) or 13vPnC/PPSV23 (712 participants); 2 participants in the 20vPnC/saline group and 2 participants in the 13vPnC/PPSV23 group were not vaccinated, therefore, a total of 1421 participants were vaccinated and included in the summary..
Groups:
- 20vPnC/Saline: Participants aged 60 years and above received a single dose of 0.5 milliliter (mL) 20vPnC intramuscularly at Vaccination 1 (Day 1) and a single dose of 0.5 mL saline intramuscularly at Vaccination 2 (28 to 42 Days after vaccination1).
- 13vPnC/PPSV23: Participants 60 years of age and above received a single dose of 0.5 mL 13vPnC intramuscularly at Vaccination 1 (Day 1) and a single dose of 0.5 mL intramuscularly PPSV23 at Vaccination 2 (28 to 42 Days after Vaccination 1).
Period: Overall Study
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Started (Participants Vaccinated with Vaccination 1) | 711 | 710
Vaccinated With Vaccination 2 | 695 | 699
Completed | 692 | 699
Not Completed | 19 | 11
Not completed — Adverse Event | 6 | 4
Not completed — Protocol Violation | 4 | 0
Not completed — Withdrawal by Subject | 8 | 5
Not completed — No longer meets eligibility criteria | 1 | 0
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who receive at least 1 dose of the study intervention (20vPnC, 13vPnC, PPSV23 or saline).
Groups:
- 20vPnC/Saline: Participants aged 60 years and above received a single dose of 0.5 mL 20vPnC intramuscularly at Vaccination 1 (Day 1) and a single dose of 0.5 mL saline intramuscularly at Vaccination 2 (28 to 42 Days after vaccination1).
- Total: Total of all reporting groups
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23 | Total
Number analyzed (Participants) | 711 | 710 | 1421
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (4.46) | 66.2 (4.83) | 66.1 (4.65)
Age, Customized [Number; unit: Participants]
  60 to 64 years | 314 | 314 | 628
  65 to 74 years | 366 | 353 | 719
  ≥75 years | 31 | 43 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 315 | 315 | 630
  Male | 396 | 395 | 791
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 711 | 710 | 1421
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 711 | 710 | 1421
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Prompted Local Reactions Within 10 Days After Vaccination 1 (20vPnC or 13vPnC)
Description: Reactions were collected in the e-diary including redness, swelling, and pain at the injection site. Exact 2-sided CI was calculated based on the Clopper and Pearson method.
  Redness and swelling were graded as mild (>2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), and severe (>10.0 cm).
  Pain at the injection site was graded as mild (does not interfere with activity), moderate (interferes with activity), and severe (prevents daily activity).
Time Frame: Within 10 days after 20vPnC in the 20vPnC/Saline group or 13vPnC in the 13vPnC/PPSV23 group
Population: Safety population included all participants who received at least 1 dose of the study intervention (20vPnC, 13vPnC, PPSV23 or saline) and had safety follow-up after any vaccination. Here, "Number of Participants Analyzed"=number of participants with any e-diary data reported after 20vPnC or 13vPnC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 710 | 710
percentage of participants
  Redness-Any | 12.4 [10.1 to 15.0] | 9.7 [7.6 to 12.1]
  Redness-Mild | 6.2 [4.5 to 8.2] | 4.5 [3.1 to 6.3]
  Redness-Moderate | 4.8 [3.3 to 6.6] | 3.9 [2.6 to 5.6]
  Redness-Severe | 1.4 [0.7 to 2.6] | 1.3 [0.6 to 2.4]
  Swelling-Any | 10.4 [8.3 to 12.9] | 7.5 [5.6 to 9.7]
  Swelling-Mild | 5.4 [3.8 to 7.3] | 3.5 [2.3 to 5.2]
  Swelling-Moderate | 4.5 [3.1 to 6.3] | 3.1 [2.0 to 4.7]
  Swelling-Severe | 0.6 [0.2 to 1.4] | 0.8 [0.3 to 1.8]
  Pain at the injection site-Any | 52.3 [48.5 to 56.0] | 50.7 [47.0 to 54.4]
  Pain at the injection site-Mild | 45.6 [41.9 to 49.4] | 46.3 [42.6 to 50.1]
  Pain at the injection site-Moderate | 6.5 [4.8 to 8.5] | 4.1 [2.8 to 5.8]
  Pain at the injection site-Severe | 0.1 [0.0 to 0.8] | 0.3 [0.0 to 1.0]

2. Primary Outcome: Percentage of Participants With Prompted Systemic Events Within 7 Days After Vaccination 1 (20vPnC or 13vPnC)
Description: Events were collected in the e-diary including fever, headache, fatigue, muscle pain, and joint pain. Exact 2-sided CI was calculated based on the Clopper and Pearson method.
  Fever was categorized as ≥38.0 degree Celsius (°C), ≥38.0°C to 38.4°C, >38.4°C to 38.9°C, >38.9°C to 40.0°C, and >40.0°C.
  Fatigue, headache, muscle pain, and joint pain were graded as mild (does not interfere with activity), moderate (some interference with activity), and severe (prevents daily activity).
Time Frame: Within 7 days after 20vPnC in the 20vPnC/Saline group or 13vPnC in the 13vPnC/PPSV23 group
Population: Safety population included all participants who received at least 1 dose of the study intervention (20vPnC, 13vPnC, PPSV23 or saline) and had safety follow-up after any vaccination. Here, "Number of Participants Analyzed" is number of participants with any e-diary data reported after 20vPnC or 13vPnC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 710 | 710
percentage of participants
  Fever ≥38.0°C | 0.1 [0.0 to 0.8] | 0.6 [0.2 to 1.4]
  Fever ≥38.0°C to 38.4°C | 0.1 [0.0 to 0.8] | 0.3 [0.0 to 1.0]
  Fever >38.4°C to 38.9°C | 0 [0.0 to 0.5] | 0.1 [0.0 to 0.8]
  Fever >38.9°C to 40.0°C | 0 [0.0 to 0.5] | 0.1 [0.0 to 0.8]
  Fever >40.0°C | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]
  Fatigue-Any | 20.7 [17.8 to 23.9] | 23.0 [19.9 to 26.2]
  Fatigue-Mild | 18.0 [15.3 to 21.1] | 18.9 [16.1 to 21.9]
  Fatigue-Moderate | 2.7 [1.6 to 4.1] | 3.8 [2.5 to 5.5]
  Fatigue-Severe | 0 [0.0 to 0.5] | 0.3 [0.0 to 1.0]
  Headache-Any | 9.2 [7.1 to 11.5] | 11.0 [8.8 to 13.5]
  Headache-Mild | 8.2 [6.3 to 10.4] | 9.6 [7.5 to 12.0]
  Headache-Moderate | 1.0 [0.4 to 2.0] | 1.1 [0.5 to 2.2]
  Headache-Severe | 0 [0.0 to 0.5] | 0.3 [0.0 to 1.0]
  Muscle pain-Any | 17.6 [14.9 to 20.6] | 17.9 [15.1 to 20.9]
  Muscle pain-Mild | 15.2 [12.6 to 18.1] | 14.8 [12.3 to 17.6]
  Muscle pain-Moderate | 2.3 [1.3 to 3.6] | 3.0 [1.8 to 4.5]
  Muscle pain-Severe | 0.1 [0.0 to 0.8] | 0.1 [0.0 to 0.8]
  Joint pain-Any | 6.8 [5.0 to 8.9] | 7.9 [6.0 to 10.1]
  Joint pain-Mild | 5.2 [3.7 to 7.1] | 5.9 [4.3 to 7.9]
  Joint pain-Moderate | 1.5 [0.8 to 2.8] | 2.0 [1.1 to 3.3]
  Joint pain-Severe | 0 [0.0 to 0.5] | 0 [0.0 to 0.5]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination 1 (20vPnC or 13vPnC)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Within 1 month after 20vPnC in the 20vPnC/Saline group or 13vPnC in the 13vPnC/PPSV23 group
Population: Safety population included all participants who received at least 1 dose of the study intervention (20vPnC, 13vPnC, PPSV23 or saline) and had safety follow-up after any vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 711 | 710
percentage of participants | 5.6 [4.0 to 7.6] | 5.9 [4.3 to 7.9]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Within 1 Month After Vaccination 1 (20vPnC or 13vPnC)
Description: An SAE was any untoward medical occurrence at any dose that resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; resulted in congenital anomaly/birth defect or that was considered to be an important medical event.
Time Frame: Within 1 Month After Vaccination 1 (20vPnC or 13vPnC)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 711 | 710
percentage of participants | 0.4 [0.1 to 1.2] | 0.6 [0.2 to 1.4]

5. Primary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for 13-matched Serotypes at 1 Month After Vaccination 1 (20vPnC or 13vPnC)
Description: OPA titers were determined for the 13 matching pneumococcal serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F. GMTs and 2-sided CIs were calculated by exponentiating the Least Square (LS) means and the corresponding CIs based on analysis of log-transformed OPA titers using a regression model with vaccine group, sex, smoking status, age at vaccination in years (continuous), baseline log-transformed OPA titers, and country.
Time Frame: 1 month after 20vPnC in the 20vPnC/Saline group or 13vPnC in the 13vPnC/PPSV23 group
Population: Participants analyzed=Evaluable 13-matched immunogenicity population (for any serotype) included participants who were enrolled, received Vaccination 1 as randomized, had at least 1 valid OPA titer for any of the 13 matched serotypes from the blood collection 27 to 49 days after Vaccination 1, had no other major protocol deviations (PDs). Number Analyzed=participants evaluable for this outcome measure (OM) at specified row.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 688 | 689
titer
  Serotype 1: number analyzed (Participants) | 687 | 688
  Serotype 1 | 207 [177 to 242] | 267 [229 to 311]
  Serotype 3: number analyzed (Participants) | 683 | 687
  Serotype 3 | 50 [45 to 55] | 56 [50 to 62]
  Serotype 4: number analyzed (Participants) | 678 | 680
  Serotype 4 | 813 [696 to 949] | 1029 [881 to 1202]
  Serotype 5: number analyzed (Participants) | 688 | 687
  Serotype 5 | 96 [82 to 112] | 125 [107 to 145]
  Serotype 6A: number analyzed (Participants) | 685 | 687
  Serotype 6A | 1286 [1088 to 1520] | 1475 [1249 to 1742]
  Serotype 6B: number analyzed (Participants) | 668 | 675
  Serotype 6B | 1399 [1196 to 1637] | 1537 [1314 to 1798]
  Serotype 7F: number analyzed (Participants) | 684 | 686
  Serotype 7F | 1735 [1578 to 1907] | 2076 [1889 to 2282]
  Serotype 9V: number analyzed (Participants) | 681 | 681
  Serotype 9V | 1467 [1285 to 1674] | 1663 [1459 to 1895]
  Serotype 14: number analyzed (Participants) | 671 | 673
  Serotype 14 | 704 [602 to 824] | 647 [554 to 756]
  Serotype 18C | 1325 [1142 to 1538] | 1826 [1575 to 2117]
  Serotype 19A: number analyzed (Participants) | 684 | 684
  Serotype 19A | 864 [750 to 994] | 1172 [1018 to 1349]
  Serotype 19F: number analyzed (Participants) | 681 | 683
  Serotype 19F | 365 [310 to 431] | 574 [487 to 676]
  Serotype 23F: number analyzed (Participants) | 688 | 687
  Serotype 23F | 290 [239 to 351] | 361 [298 to 437]
Statistical Analysis 1: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 1: the ratio of GMT (GMR) (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — Noninferiority for a serotype was declared if the lower bound of the 2-sided 95% CI for the ratio of GMT20vPnC/saline to GMT13vPnC/PPSV23 for that serotype is greater than 0.5 (2-fold criterion); Ratio of GMTs (20vPnC/13vPnC) = 0.78, 95% CI 2-sided [0.66 to 0.92]
Statistical Analysis 2: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 3: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/13vPnC) = 0.89, 95% CI 2-sided [0.79 to 0.99]
Statistical Analysis 3: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 4: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/13vPnC) = 0.79, 95% CI 2-sided [0.67 to 0.94]
Statistical Analysis 4: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 5: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/13vPnC) = 0.77, 95% CI 2-sided [0.65 to 0.91]
Statistical Analysis 5: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 6A: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/13vPnC) = 0.87, 95% CI 2-sided [0.73 to 1.05]
Statistical Analysis 6: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 6B: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/13vPnC) = 0.91, 95% CI 2-sided [0.77 to 1.08]
Statistical Analysis 7: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 7F: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/13vPnC) = 0.84, 95% CI 2-sided [0.75 to 0.93]
Statistical Analysis 8: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 9V: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/13vPnC) = 0.88, 95% CI 2-sided [0.76 to 1.02]
Statistical Analysis 9: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 14: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/13vPnC) = 1.09, 95% CI 2-sided [0.92 to 1.29]
Statistical Analysis 10: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 18C: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/13vPnC) = 0.73, 95% CI 2-sided [0.62 to 0.85]
Statistical Analysis 11: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 19A: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/13vPnC) = 0.74, 95% CI 2-sided [0.63 to 0.86]
Statistical Analysis 12: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 19F: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/13vPnC) = 0.64, 95% CI 2-sided [0.53 to 0.76]
Statistical Analysis 13: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 23F: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/13vPnC) = 0.80, 95% CI 2-sided [0.65 to 0.99]

6. Primary Outcome: Pneumococcal OPA GMTs for 7 Additional Serotypes at 1 Month After Vaccination 1 (20vPnC) or 1 Month After Vaccination 2 (PPSV23)
Description: OPA titers were determined for serotypes: 8, 10A, 11A, 12F, 15B, 22F, and 33F. GMTs and 2-sided CIs were calculated by exponentiating the LS means and the corresponding CIs based on analysis of log-transformed OPA titers using a regression model with vaccine group, sex, smoking status, age at vaccination in years (continuous), baseline log-transformed OPA titers, and country.
Time Frame: 1 month after 20vPnC in the 20vPnC/Saline group or 1 month after PPSV23 in the 13vPnC/PPSV23 group.
Population: Participants Analyzed=Evaluable 7-additional immunogenicity population (for any serotype) included participants who were enrolled, received 20vPnC in the 20vPnC/saline group or received both vaccinations in the 13vPnC/PPSV23 group, had at least 1 valid OPA titers for any of the 7 additional serotypes from the blood collection 27 to 49 days after Vaccination 1 or 2 respectively, had no other major PDs. Number Analyzed=participants evaluable for this OM at specified row.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 689 | 693
titer
  Serotype 8: number analyzed (Participants) | 669 | 674
  Serotype 8 | 561 [490 to 642] | 971 [850 to 1110]
  Serotype 10A: number analyzed (Participants) | 664 | 663
  Serotype 10A | 1661 [1422 to 1939] | 777 [667 to 906]
  Serotype 11A: number analyzed (Participants) | 652 | 639
  Serotype 11A | 3331 [2834 to 3913] | 1933 [1644 to 2274]
  Serotype 12F: number analyzed (Participants) | 647 | 638
  Serotype 12F | 3543 [2976 to 4217] | 2104 [1766 to 2507]
  Serotype 15B: number analyzed (Participants) | 652 | 651
  Serotype 15B | 1265 [1039 to 1539] | 593 [487 to 723]
  Serotype 22F: number analyzed (Participants) | 657 | 656
  Serotype 22F | 2818 [2345 to 3388] | 1737 [1445 to 2089]
  Serotype 33F: number analyzed (Participants) | 660 | 653
  Serotype 33F | 6675 [5751 to 7748] | 5853 [5046 to 6788]
Statistical Analysis 1: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 8: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/PPSV23) = 0.58, 95% CI 2-sided [0.50 to 0.67]
Statistical Analysis 2: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 10A: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/PPSV23) = 2.14, 95% CI 2-sided [1.80 to 2.53]
Statistical Analysis 3: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 11A: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/PPSV23) = 1.72, 95% CI 2-sided [1.44 to 2.06]
Statistical Analysis 4: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 12F: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/PPSV23) = 1.68, 95% CI 2-sided [1.39 to 2.04]
Statistical Analysis 5: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 15B: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/PPSV23) = 2.13, 95% CI 2-sided [1.72 to 2.64]
Statistical Analysis 6: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 22F: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/PPSV23) = 1.62, 95% CI 2-sided [1.33 to 1.98]
Statistical Analysis 7: Comparison: 20vPnC/Saline vs 13vPnC/PPSV23; Serotype 33F: GMR (the 20vPnC/saline group to the 13vPnC/PPSV23 group) and the 2-sided 95% CI; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Ratio of GMTs (20vPnC/PPSV23) = 1.14, 95% CI 2-sided [0.97 to 1.34]

7. Secondary Outcome: OPA Geometric Mean Fold Rise (GMFRs) For 13-matched Serotypes From Before To 1 Month After Vaccination 1 (20vPnC or 13vPnC)
Description: GMFRs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding CIs (based on the Student's t distribution), for serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: Before Vaccination 1 to 1 month after 20vPnC in the 20vPnC/saline group or 13vPnC in the 13vPnC/PPSV23 group.
Population: Participants Analyzed=Evaluable 13-matched immunogenicity population (for any serotype) included participants who were enrolled, received Vaccination 1 as randomized, had at least 1 valid OPA titer for any of the 13 matched serotypes from the blood collection 27 to 49 days after Vaccination 1, had no other major PDs. Number analyzed in each row=participants evaluable with OPA titers available at both timepoints at specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 688 | 689
fold rise
  Serotype 1: number analyzed (Participants) | 685 | 686
  Serotype 1 | 13.1 [11.5 to 14.9] | 16.3 [14.2 to 18.7]
  Serotype 3: number analyzed (Participants) | 680 | 679
  Serotype 3 | 4.8 [4.4 to 5.3] | 5.4 [4.9 to 5.9]
  Serotype 4: number analyzed (Participants) | 648 | 661
  Serotype 4 | 30.1 [26.0 to 34.9] | 35.7 [30.5 to 41.7]
  Serotype 5: number analyzed (Participants) | 685 | 685
  Serotype 5 | 5.4 [4.8 to 6.0] | 6.9 [6.1 to 7.8]
  Serotype 6A: number analyzed (Participants) | 672 | 674
  Serotype 6A | 24.3 [20.9 to 28.3] | 26.9 [23.0 to 31.6]
  Serotype 6B: number analyzed (Participants) | 635 | 637
  Serotype 6B | 14.8 [12.8 to 17.3] | 15.7 [13.5 to 18.4]
  Serotype 7F: number analyzed (Participants) | 639 | 636
  Serotype 7F | 5.9 [5.3 to 6.6] | 7.0 [6.3 to 7.9]
  Serotype 9V: number analyzed (Participants) | 646 | 667
  Serotype 9V | 7.1 [6.3 to 8.0] | 7.5 [6.6 to 8.5]
  Serotype 14: number analyzed (Participants) | 649 | 659
  Serotype 14 | 8.7 [7.6 to 10.0] | 7.8 [6.7 to 9.0]
  Serotype 18C: number analyzed (Participants) | 678 | 684
  Serotype 18C | 18.6 [16.0 to 21.5] | 24.6 [21.3 to 28.5]
  Serotype 19A: number analyzed (Participants) | 675 | 675
  Serotype 19A | 24.1 [20.9 to 27.8] | 30.2 [26.2 to 34.8]
  Serotype 19F: number analyzed (Participants) | 674 | 675
  Serotype 19F | 8.9 [7.8 to 10.2] | 13.5 [11.7 to 15.6]
  Serotype 23F: number analyzed (Participants) | 685 | 684
  Serotype 23F | 18.7 [15.9 to 22.0] | 22.2 [18.8 to 26.2]

8. Secondary Outcome: OPA GMFRs for 7 Additional Serotypes From Before to 1 Month After Vaccination 1 (20vPnC) or From Before Vaccination 1 to 1 Month After Vaccination 2 (PPSV23)
Description: GMFRs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding CIs (based on the Student's t distribution), for serotypes 8, 10A, 11A, 12F, 15B, 22F, and 33F.
Time Frame: From before Vaccination 1 (20vPnC) to 1 month after Vaccination 1 (20vPnC) in the 20vPnC/Saline group or from before Vaccination 1 (13vPnC) to 1 month after Vaccination 2 (PPSV23) in the 13vPnC/PPSV23 group
Population: Participants Analyzed=Evaluable 7-additional immunogenicity population (for any serotype) included participants who were enrolled, received 20vPnC in the 20vPnC/saline group or received both vaccinations in the 13vPnC/PPSV23 group, had ≥1 valid OPA titers for any of the 7 additional serotypes from the blood collection 27-49 days after Vaccination 1 or 2 respectively, had no other major PDs.Number Analyzed=participants evaluable with OPA titers available at both timepoints at specified serotypes
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 689 | 693
fold rise
  Serotype 8: number analyzed (Participants) | 661 | 665
  Serotype 8 | 17.9 [15.7 to 20.3] | 30.2 [26.5 to 34.4]
  Serotype 10A: number analyzed (Participants) | 638 | 633
  Serotype 10A | 13.1 [11.4 to 15.1] | 6.1 [5.4 to 7.0]
  Serotype 11A: number analyzed (Participants) | 563 | 552
  Serotype 11A | 14.5 [12.2 to 17.1] | 7.3 [6.2 to 8.5]
  Serotype 12F: number analyzed (Participants) | 620 | 602
  Serotype 12F | 69.1 [58.9 to 81.1] | 38.2 [32.2 to 45.3]
  Serotype 15B: number analyzed (Participants) | 637 | 632
  Serotype 15B | 25.9 [21.7 to 31.0] | 11.8 [10.0 to 14.0]
  Serotype 22F: number analyzed (Participants) | 612 | 610
  Serotype 22F | 41.1 [33.4 to 50.5] | 23.1 [19.2 to 27.9]
  Serotype 33F: number analyzed (Participants) | 640 | 623
  Serotype 33F | 7.5 [6.5 to 8.5] | 6.2 [5.5 to 7.1]

9. Secondary Outcome: Percentage of Participants With ≥4 Fold Rise for 13-matched Serotypes of OPA Titers From Before to 1 Month After Vaccination 1 (20vPnC or 13vPnC)
Description: The percentage of participants with a ≥4-fold rise in OPA titers and associated 95% CI before vaccination to 1 month after vaccination with 20vPnC or 13vPnC for the 13 matching serotypes, including 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F were summarized.
Time Frame: From before Vaccination 1 to 1 month after 20vPnC in the 20vPnC/Saline group or 13vPnC in the 13vPnC/PPSV23 group
Population: Participants Analyzed=Evaluable 13-matched immunogenicity population (for any serotype) included participants who were enrolled, received Vaccination 1 as randomized, had at least 1 valid OPA titer for any of the 13 matched serotypes from the blood collection 27 to 49 days after Vaccination 1, had no other major PDs. Number Analyzed=participants evaluable with OPA titers available at both timepoints at specified serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 688 | 689
percentage of participants
  Serotype 1: number analyzed (Participants) | 685 | 686
  Serotype 1 | 72.6 [69.0 to 75.9] | 74.2 [70.8 to 77.4]
  Serotype 3: number analyzed (Participants) | 680 | 679
  Serotype 3 | 57.6 [53.8 to 61.4] | 59.4 [55.5 to 63.1]
  Serotype 4: number analyzed (Participants) | 648 | 661
  Serotype 4 | 80.1 [76.8 to 83.1] | 79.6 [76.3 to 82.6]
  Serotype 5: number analyzed (Participants) | 685 | 685
  Serotype 5 | 54.9 [51.1 to 58.7] | 59.6 [55.8 to 63.3]
  Serotype 6A: number analyzed (Participants) | 672 | 674
  Serotype 6A | 78.9 [75.6 to 81.9] | 77.6 [74.3 to 80.7]
  Serotype 6B: number analyzed (Participants) | 635 | 637
  Serotype 6B | 71.2 [67.5 to 74.7] | 70.6 [66.9 to 74.2]
  Serotype 7F: number analyzed (Participants) | 639 | 636
  Serotype 7F | 55.7 [51.8 to 59.6] | 61.9 [58.0 to 65.7]
  Serotype 9V: number analyzed (Participants) | 646 | 667
  Serotype 9V | 60.5 [56.6 to 64.3] | 62.8 [59.0 to 66.5]
  Serotype 14: number analyzed (Participants) | 649 | 659
  Serotype 14 | 59.5 [55.6 to 63.3] | 53.4 [49.5 to 57.3]
  Serotype 18C: number analyzed (Participants) | 678 | 684
  Serotype 18C | 73.3 [69.8 to 76.6] | 79.1 [75.9 to 82.1]
  Serotype 19A: number analyzed (Participants) | 675 | 675
  Serotype 19A | 79.6 [76.3 to 82.5] | 82.4 [79.3 to 85.2]
  Serotype 19F: number analyzed (Participants) | 674 | 675
  Serotype 19F | 62.5 [58.7 to 66.1] | 69.9 [66.3 to 73.4]
  Serotype 23F: number analyzed (Participants) | 685 | 684
  Serotype 23F | 69.8 [66.2 to 73.2] | 72.5 [69.0 to 75.8]

10. Secondary Outcome: Percentage of Participants With ≥4 Fold Rise in 7 Additional Serotypes of OPA Titers From Before Vaccination 1 to 1 Month After Vaccination 1 (20vPnC) or From Before Vaccination 1 to 1 Month After Vaccination 2 (PPSV23)
Description: The percentage of participants with a ≥4-fold rise in OPA titers and associated 95% CI before vaccination to 1 month after vaccination with 20vPnC or PPSV23 for the 7 additional serotypes, including 8, 10A, 11A, 12F, 15B, 22F, and 33F were summarized.
Time Frame: as for outcome 8
Population: Participants Analyzed=Evaluable 7-additional immunogenicity population (for any serotype): participants who were enrolled, received 20vPnC in the 20vPnC/saline group or received both vaccinations in the 13vPnC/PPSV23 group, had at least 1 valid OPA titers for any of the 7 additional serotypes from the blood collection 27 to 49 days after Vaccination 1 or 2 respectively, had no other major PDs. Number Analyzed=participants evaluable with OPA titers available at both timepoints at specified rows
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 689 | 693
percentage of participants
  Serotype 8: number analyzed (Participants) | 661 | 665
  Serotype 8 | 80.5 [77.3 to 83.4] | 86.3 [83.5 to 88.8]
  Serotype 10A: number analyzed (Participants) | 638 | 633
  Serotype 10A | 70.2 [66.5 to 73.7] | 56.1 [52.1 to 60.0]
  Serotype 11A: number analyzed (Participants) | 563 | 552
  Serotype 11A | 69.4 [65.5 to 73.2] | 53.1 [48.8 to 57.3]
  Serotype 12F: number analyzed (Participants) | 620 | 602
  Serotype 12F | 86.9 [84.0 to 89.5] | 80.7 [77.3 to 83.8]
  Serotype 15B: number analyzed (Participants) | 637 | 632
  Serotype 15B | 73.6 [70.0 to 77.0] | 59.7 [55.7 to 63.5]
  Serotype 22F: number analyzed (Participants) | 612 | 610
  Serotype 22F | 75.5 [71.9 to 78.8] | 70.8 [67.0 to 74.4]
  Serotype 33F: number analyzed (Participants) | 640 | 623
  Serotype 33F | 61.1 [57.2 to 64.9] | 58.1 [54.1 to 62.0]

11. Secondary Outcome: Percentage of Participants With 13-matched Serotypes of OPA Titers ≥The Lower Limit of Quantitation (LLOQ) 1 Month After Vaccination 1 (20vPnC or 13vPnC)
Description: The percentage of participants with OPA titers ≥LLOQ and associated 95% CIs were calculated for the time point 1 month after vaccination with 20vPnC or 13vPnC for serotypes: 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F.
Time Frame: 1 month after 20vPnC in the 20vPnC/saline group or 13vPnC in the 13vPnC/PPSV23 group
Population: Participants Analyzed=Evaluable 13-matched immunogenicity population (for any serotype) included participants who were enrolled, received Vaccination 1 as randomized, had at least 1 valid OPA titer for any of the 13 matched serotypes from the blood collection 27 to 49 days after Vaccination 1, had no other major PDs. Number analyzed=participants evaluable for this OM at specified rows.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 688 | 689
percentage of participants
  Serotype 1: number analyzed (Participants) | 687 | 688
  Serotype 1 | 84.3 [81.3 to 86.9] | 85.6 [82.8 to 88.1]
  Serotype 3: number analyzed (Participants) | 683 | 687
  Serotype 3 | 82.3 [79.2 to 85.1] | 82.4 [79.3 to 85.2]
  Serotype 4: number analyzed (Participants) | 678 | 680
  Serotype 4 | 91.7 [89.4 to 93.7] | 92.4 [90.1 to 94.2]
  Serotype 5: number analyzed (Participants) | 688 | 687
  Serotype 5 | 67.6 [63.9 to 71.1] | 70.7 [67.2 to 74.1]
  Serotype 6A: number analyzed (Participants) | 685 | 687
  Serotype 6A | 89.8 [87.3 to 91.9] | 88.8 [86.2 to 91.1]
  Serotype 6B: number analyzed (Participants) | 668 | 675
  Serotype 6B | 91.5 [89.1 to 93.5] | 90.2 [87.7 to 92.4]
  Serotype 7F: number analyzed (Participants) | 684 | 686
  Serotype 7F | 98.1 [96.8 to 99.0] | 98.0 [96.6 to 98.9]
  Serotype 9V: number analyzed (Participants) | 681 | 681
  Serotype 9V | 87.2 [84.5 to 89.6] | 88.3 [85.6 to 90.6]
  Serotype 14: number analyzed (Participants) | 671 | 673
  Serotype 14 | 92.1 [89.8 to 94.0] | 88.4 [85.7 to 90.7]
  Serotype 18C | 93.3 [91.2 to 95.1] | 94.8 [92.8 to 96.3]
  Serotype 19A: number analyzed (Participants) | 684 | 684
  Serotype 19A | 95.0 [93.1 to 96.5] | 96.8 [95.2 to 98.0]
  Serotype 19F: number analyzed (Participants) | 681 | 683
  Serotype 19F | 76.4 [73.0 to 79.5] | 82.3 [79.2 to 85.1]
  Serotype 23F: number analyzed (Participants) | 688 | 687
  Serotype 23F | 79.8 [76.6 to 82.7] | 82.4 [79.3 to 85.2]

12. Secondary Outcome: Percentage of Participants With Pneumococcal OPA Titers ≥LLOQ for the 7 Additional Serotypes at 1 Month After Vaccination 1 (20vPnC) or 1 Month After Vaccination 2 (PPSV23)
Description: The percentage of participants with OPA titers ≥LLOQ and associated 95% CIs were calculated for the time point 1 month after vaccination with 20vPnC in the 20vPnC/saline groups or PPSV23 in the 13vPnC/PPSV23 group for serotypes: 8, 10A, 11A, 12F, 15B, 22F, and 33F.
Time Frame: 1 month after Vaccination 1 (20vPnC) in the 20vPnC/saline group or a month after Vaccination 2 (PPSV23) in the 13vPnC/PPSV23 group
Population: Participants Analyzed=Evaluable 7-additional immunogenicity population (for any serotype): participants who were enrolled, received 20vPnC if randomized to 20vPnC/saline group or received both vaccinations if randomized to 13vPnC/PPSV23 group, had at least 1 valid OPA titers for any of the 7 additional serotypes from the blood collection 27 to 49 days after Vaccination 1 or Vaccination 2 respectively, had no other major PDs. Number analyzed=participants evaluable at specified rows.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 689 | 693
percentage of participants
  Serotype 8: number analyzed (Participants) | 669 | 674
  Serotype 8 | 95.2 [93.3 to 96.7] | 96.7 [95.1 to 97.9]
  Serotype 10A: number analyzed (Participants) | 664 | 663
  Serotype 10A | 91.1 [88.7 to 93.2] | 82.1 [78.9 to 84.9]
  Serotype 11A: number analyzed (Participants) | 652 | 639
  Serotype 11A | 96.9 [95.3 to 98.1] | 92.3 [90.0 to 94.3]
  Serotype 12F: number analyzed (Participants) | 647 | 638
  Serotype 12F | 96.9 [95.3 to 98.1] | 91.7 [89.3 to 93.7]
  Serotype 15B: number analyzed (Participants) | 652 | 651
  Serotype 15B | 90.2 [87.6 to 92.4] | 80.3 [77.1 to 83.3]
  Serotype 22F: number analyzed (Participants) | 657 | 656
  Serotype 22F | 96.5 [94.8 to 97.8] | 93.3 [91.1 to 95.1]
  Serotype 33F: number analyzed (Participants) | 660 | 653
  Serotype 33F | 97.4 [95.9 to 98.5] | 96.5 [94.8 to 97.8]

13. Secondary Outcome: Percentage of Participants With Prompted Local Reactions Within 10 Days After Vaccination 2 (PPSV23 or Saline) in Participants Enrolled at Japan Sites
Description: Reactions within 10 days after Vaccination 2 (PPSV23 or saline) in participants enrolled at Japan sites were collected in the e-diary including redness, swelling, and pain at the injection site. Exact 2-sided CI was calculated based on the Clopper and Pearson method.
  Redness and swelling were graded as mild (>2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm), and severe (>10.0 cm).
  Pain at the injection site was grades as mild (does not interfere with activity), moderate (interferes with activity), and severe (prevents daily activity).
  This endpoint was requested by local Japan regulator.
Time Frame: Within 10 days after saline in 20vPnC/Saline group or PPSV23 in 13vPnC/PPSV23 group
Population: Safety population included all participants enrolled at Japan sites who received at least 1 dose of the study intervention (20vPnC, 13vPnC, PPSV23 or saline) and had safety follow-up after any vaccination. Here, "Number of Participants Analyzed" is participants enrolled at Japan sites with any e-diary data reported after PPSV23 or saline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 409 | 413
percentage of participants
  Redness-Any | 1.2 [0.4 to 2.8] | 17.2 [13.7 to 21.2]
  Redness-Mild | 1.2 [0.4 to 2.8] | 3.6 [2.0 to 5.9]
  Redness-Moderate | 0 [0 to 0.9] | 8.2 [5.8 to 11.3]
  Redness-Severe | 0 [0 to 0.9] | 5.3 [3.4 to 8.0]
  Swelling-Any | 1.0 [0.3 to 2.5] | 28.3 [24.0 to 32.9]
  Swelling-Mild | 1.0 [0.3 to 2.5] | 7.7 [5.4 to 10.8]
  Swelling-Moderate | 0 [0 to 0.9] | 13.6 [10.4 to 17.2]
  Swelling-Severe | 0 [0 to 0.9] | 7.0 [4.8 to 9.9]
  Pain at the injection site-Any | 5.6 [3.6 to 8.3] | 73.1 [68.6 to 77.3]
  Pain at the injection site-Mild | 5.6 [3.6 to 8.3] | 46.0 [41.1 to 50.9]
  Pain at the injection site-Moderate | 0 [0.0 to 0.9] | 24.5 [20.4 to 28.9]
  Pain at the injection site-Severe | 0 [0.0 to 0.9] | 2.7 [1.3 to 4.7]

14. Secondary Outcome: Percentage of Participants With Prompted Systemic Events Within 7 Days After Vaccination 2 (PPSV23 or Saline) in Participants Enrolled at Japan Sites
Description: Events within 7 days after Vaccination 2 (PPSV23 or saline) in participants enrolled at Japan sites were collected in the e-diary including fever, headache, fatigue, muscle pain, and joint pain. Exact 2-sided CI was calculated based on the Clopper and Pearson method.
  Fever was categorized as ≥38.0 °C, ≥38.0°C to 38.4°C, >38.4°C to 38.9°C, >38.9°C to 40.0°C, and >40.0°C.
  Fatigue, headache, muscle pain, and joint pain were grades as mild (does not interfere with activity), moderate (some interference with activity), and severe (prevents daily activity).
  This endpoint was requested by local Japan regulator.
Time Frame: Within 7 days after saline in 20vPnC/Saline group or PPSV23 in 13vPnC/PPSV23 group
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC/Saline | 13vPnC/PPSV23
Number analyzed (Participants) | 409 | 413
percentage of participants
  Fever ≥38.0°C | 0.2 [0.0 to 1.4] | 1.7 [0.7 to 3.5]
  Fever ≥38.0°C to 38.4°C | 0 [0.0 to 0.9] | 1.5 [0.5 to 3.1]
  Fever >38.4°C to 38.9°C | 0.2 [0.0 to 1.4] | 0.2 [0.0 to 1.3]
  Fever >38.9°C to 40.0°C | 0 [0.0 to 0.9] | 0 [0.0 to 0.9]
  Fever >40.0°C | 0 [0.0 to 0.9] | 0 [0.0 to 0.9]
  Fatigue-Any | 9.5 [6.9 to 12.8] | 22.5 [18.6 to 26.9]
  Fatigue-Mild | 7.8 [5.4 to 10.9] | 15.7 [12.4 to 19.6]
  Fatigue-Moderate | 1.5 [0.5 to 3.2] | 6.1 [4.0 to 8.8]
  Fatigue-Severe | 0.2 [0.0 to 1.4] | 0.7 [0.2 to 2.1]
  Headache-Any | 4.9 [3.0 to 7.5] | 9.4 [6.8 to 12.7]
  Headache-Mild | 4.4 [2.6 to 6.9] | 8.0 [5.6 to 11.0]
  Headache-Moderate | 0.5 [0.1 to 1.8] | 1.2 [0.4 to 2.8]
  Headache-Severe | 0 [0.0 to 0.9] | 0.2 [0.0 to 1.3]
  Muscle pain-Any | 4.2 [2.4 to 6.6] | 25.4 [21.3 to 29.9]
  Muscle pain-Mild | 3.7 [2.1 to 6.0] | 16.5 [13.0 to 20.4]
  Muscle pain-Moderate | 0.5 [0.1 to 1.8] | 8.0 [5.6 to 11.0]
  Muscle pain-Severe | 0 [0.0 to 0.9] | 1.0 [0.3 to 2.5]
  Joint pain-Any | 1.7 [0.7 to 3.5] | 6.1 [4.0 to 8.8]
  Joint pain-Mild | 1.5 [0.5 to 3.2] | 4.4 [2.6 to 6.8]
  Joint pain-Moderate | 0.2 [0.0 to 1.4] | 1.5 [0.5 to 3.1]
  Joint pain-Severe | 0 [0.0 to 0.9] | 0.2 [0.0 to 1.3]

ADVERSE EVENTS:
Time Frame: SAEs, non-serious AEs (NSAEs), and deaths were reported from Vaccination 1 (Day 1) to 28-42 days after Vaccination 1 and Vaccination 2 to 28-42 days after Vaccination 2 from all participants. The e-diary was collected 10 days for local reactions and 7 days for systemic events after Vaccination 1 for all participants, and after Vaccination 2 for Japan participants only.
Description: Same event may appear as NSAE and SAE, what is presented are distinct events. Event may be categorized as SAE in 1 participant and as NSAE in another participant or 1 participant may have experienced both SAE and NSAE during study. Participants received 20vPnC followed by saline in the 20vPnC/saline group or 13vPnC followed by PPSV23 in the 13vPnC/PPSV23 group. Results were summarized by the 1-month time period following vaccination 1 or vaccination 2 for each group using the safety population.
Groups:
- 20vPnC/Saline (Vaccination 1): Participants aged 60 years and above received a single dose of 0.5 mL 20vPnC intramuscularly at Vaccination 1 (Day 1)
- 13vPnC/PPSV23 (Vaccination 1): Participants aged 60 years and above received a single dose of 0.5 mL 13vPnC intramuscularly at Vaccination 1 (Day 1).
- 20vPnC/Saline (Vaccination 2): Participants aged 60 years and above received a single dose of 0.5 mL saline intramuscularly at Vaccination 2 (28 to 42 Days after vaccination1).
- 13vPnC/PPSV23 (Vaccination 2): Participants aged 60 years and above received a single dose of 0.5mL PPSV23 intramuscularly at Vaccination 2 (28 to 42 Days after Vaccination 1).
Arm/Group | 20vPnC/Saline (Vaccination 1) | 13vPnC/PPSV23 (Vaccination 1) | 20vPnC/Saline (Vaccination 2) | 13vPnC/PPSV23 (Vaccination 2)
All-Cause Mortality (participants affected / at risk) | 0/711 | 0/710 | 0/695 | 0/699
Serious Adverse Events (participants affected / at risk) | 3/711 | 4/710 | 4/695 | 3/699
Other Adverse Events (participants affected / at risk) | 448/711 | 439/710 | 78/695 | 333/699
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20vPnC/Saline (Vaccination 1) (N=711) | 13vPnC/PPSV23 (Vaccination 1) (N=710) | 20vPnC/Saline (Vaccination 2) (N=695) | 13vPnC/PPSV23 (Vaccination 2) (N=699)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 1 | 2 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Viral rash (Infections and infestations) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 20vPnC/Saline (Vaccination 1) (N=711) | 13vPnC/PPSV23 (Vaccination 1) (N=710) | 20vPnC/Saline (Vaccination 2) (N=695) | 13vPnC/PPSV23 (Vaccination 2) (N=699)
Fatigue (FATIGUE) (General disorders) | 147 | 163 | 39 | 93
Injection site erythema (REDNESS) (General disorders) | 88 | 69 | 5 | 71
Injection site pain (PAIN) (General disorders) | 371 | 360 | 23 | 302
Injection site swelling (SWELLING) (General disorders) | 74 | 53 | 4 | 117
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 48 | 56 | 0 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 125 | 127 | 17 | 105
Headache (HEADACHE) (Nervous system disorders) | 65 | 78 | 20 | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT04875533/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT04875533/SAP_001.pdf